CLINICAL TRIAL: NCT00589472
Title: Neoadjuvant Androgen Depletion in Combination With Vorinostat Followed by Radical Prostatectomy for Localized Prostate Cancer: Total Androgen-Receptor Gene Expression Targeted Therapy (TARGET)
Brief Title: Androgen Deprivation Therapy and Vorinostat Followed by Radical Prostatectomy in Treating Patients With Localized Prostate Cancer
Acronym: TARGET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00238; NCI-2009-00238 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 06-160; MSKCC IRB 06-160; MSKCC-06160; CDR0000579559; 06-160 (Other: Memorial Sloan-Kettering Cancer Center); 7864 (Other: CTEP); N01CM62205 (NIH); N01CM62206 (NIH); P30CA008748 (NIH)
Record Dates: First submitted 2007-12-20; First posted 2008-01-09 (Estimated); Results first posted 2017-10-06 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-09

CONDITIONS: Prostate Adenocarcinoma; Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer; Stage III Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Goserelin; Leuprolide; luprolide acetate gel depot; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Antihormone therapy and enzyme inhibitor therapy) (Experimental): Patients receive bicalutamide PO QD for 1 month and leuprolide acetate IM or goserelin acetate SC once a month until surgery. Patients also receive vorinostat PO QD beginning on the first day of androgen depletion therapy and continuing for up to 8 weeks or until the day of surgery. Patients then undergo an open or laparoscopic radical prostatectomy. Patients with positive surgical margins undergo immediate adjuvant external beam radiotherapy to the prostatic fossa, based on the judgment of the treating physician.
  Interventions: Drug: Bicalutamide; Drug: Goserelin Acetate; Other: Laboratory Biomarker Analysis; Drug: Leuprolide Acetate; Procedure: Therapeutic Conventional Surgery; Drug: Vorinostat

INTERVENTIONS:
Drug: Bicalutamide — Given PO
  Other Names: Casodex; Cosudex; ICI 176,334; ICI 176334
Drug: Goserelin Acetate — Given SC
  Other Names: ZDX; Zoladex
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Leuprolide Acetate — Given IM
  Other Names: A-43818; Abbott 43818; Abbott-43818; Carcinil; Depo-Eligard; Eligard; Enanton; Enantone; Enantone-Gyn; Ginecrin; LEUP; Leuplin; Leuprorelin Acetate; Lucrin; Lucrin Depot; Lupron; Lupron Depot; Lupron Depot-3 Month; Lupron Depot-4 Month; Lupron Depot-Ped; Procren; Procrin; Prostap; TAP-144; Trenantone; Uno-Enantone; Viadur
Procedure: Therapeutic Conventional Surgery — Undergo radical prostatectomy
Drug: Vorinostat — Given PO
  Other Names: L-001079038; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza

SUMMARY:
This phase II trial studies how well androgen deprivation therapy and vorinostat followed by radical prostatectomy works in treating patients with prostate cancer that has not spread to other parts of the body. Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as bicalutamide, goserelin acetate, and leuprolide acetate, may lessen the amount of androgens made by the body. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving androgen deprivation therapy and vorinostat before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the rate of pathologic complete response in patients with localized prostate cancer treated with androgen depletion therapy (ADT) and oral vorinostat administered for a minimum of 6 weeks and maximum of 8 weeks before radical prostatectomy.

SECONDARY OBJECTIVES:

I. To determine and evaluate pre- and post-treatment levels of prostate-specific antigen (PSA), testosterone, dihydrotestosterone (DHT), dehydroepiandrosterone (DHEA), and dehydroepiandrosterone-dulfate (DHEA-S) in blood.

II. To determine and evaluate pre- and post-treatment levels of testosterone, androstenedione, androstenediol, DHT, DHEA, and DHEA-S in prostate.

III. To determine and evaluate gene and protein expression analysis including androgen receptor (AR) target genes, PSA and TMPRSS2 (transmembrane protease, serine 2), in pre-treatment biopsy and post-treatment radical prostatectomy.

IV. To determine and evaluate exploratory gene microarray analysis. V. To determine and evaluate the safety and tolerability of ADT in combination with vorinostat (SAHA) as assessed by physical examinations, adverse events, and laboratory assessments.

OUTLINE:

Patients receive bicalutamide orally (PO) once daily (QD) for 1 month and leuprolide acetate intramuscularly (IM) or goserelin acetate subcutaneously (SC) once a month until surgery. Patients also receive vorinostat PO QD beginning on the first day of androgen depletion therapy and continuing for up to 8 weeks or until the day of surgery. Patients then undergo an open or laparoscopic radical prostatectomy. Patients with positive surgical margins undergo immediate adjuvant external beam radiotherapy to the prostatic fossa, based on the judgment of the treating physician.

After completion of study treatment, patients are followed every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of prostatic adenocarcinoma in 3 or more biopsy cores, of which at least 1 core demonstrates > 30% involvement with tumor; confirmation of localized disease by magnetic resonance imaging (MRI) with endorectal probe if available
* No evidence of distant disease on a:

  * Computed tomography (CT) or MRI of the abdomen and pelvis
  * Radionuclide bone scan (with plain film or MRI confirmation as clinically indicated)
* Appropriate candidate for radical prostatectomy

  * Adequate cardiac function (evidence of cardiac disease should be evaluated to determine appropriateness of patient as a surgical candidate)
  * Candidates may have a history of deep vein thrombosis, pulmonary embolism, and/or cerebrovascular accident, or require concomitant systemic anticoagulation, if otherwise deemed to be suitable for radical prostatectomy
* White blood cell (WBC) > 3000/uL
* Platelets > 150,000/uL
* Creatinine < 2 mg/dL
* Serum PSA < 100 ng/mL
* Bilirubin < 1.5 X ULN (institutional upper limits of normal)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 2 X ULN
* Karnofsky performance status > 70%
* Willingness to undergo pretreatment transrectal ultrasound-guided prostate needle biopsy (optional)
* Willingness to use adequate contraceptive methods during study therapy and for at least 3 months after completion of therapy
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Evidence of small-cell, transitional-cell, or neuroendocrine pathologic features
* Prior hormonal therapy with (e.g. 5-alpha-reductase inhibitors, gonadotropin hormone releasing analogs, steroids, megestrol acetate, or nonstudy-related antiandrogens), chemotherapy, or herbal medications administered with the intent to treat the patient's malignancy

  * Patients on valproic acid (a histone-deacetylase inhibitor) to treat prostate cancer are not eligible
* History of allergic reactions attributed to compounds of similar chemical or biological composition to vorinostat
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would compromise compliance with study requirements
* Currently active secondary malignancy (as determined by the treating physician) other than non-melanoma skin cancer

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Slovin, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (15):
- United States (15):
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - UMDNJ - New Jersey Medical School, Newark, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - M D Anderson Cancer Center, Houston, Texas
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Antihormone Therapy and Enzyme Inhibitor Therapy)
Started | 19
Completed | 18
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Antihormone Therapy and Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response at the Time of Surgery
Description: The primary endpoint will be pathologic complete response at the time of surgery. This represents the proportion of patients with no evidence of disease in the prostate (ie, the absence of tumor in the posttherapy pathology specimen) at the time of radical prostatectomy. Pathologic complete response at the time of surgery is the primary endpoint for this study. A Simon 2-stage optimal design that differentiates between response probabilities of 0.05 and 0.20 will be used in the analysis of the pathological complete response at 12 weeks (Type I error 10% and power 90%). A maximum of 38 pts were planned for accrual onto this study. If zero or one response was observed, then the trial was to be stopped. The design had power 0.90 for a population response proportion to 0.20 using a one-sided 0.10 size test. pT2 indicates that the cancer is confined to the prostate, while pT3 indicates that there is an extraprostatic extension of the cancer.
Time Frame: At 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Antihormone Therapy and Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 18
Participants
  pT2 | 10
  pT3 | 8
  Complete Response | 0

2. Secondary Outcome: Gleason Score
Description: A Gleason score is the sum of two numbers. Pathologist determines where the cancer is most prominent and assigns the primary grade, the secondary grade is assigned based on where the cancer is next most prominent. A score from one to five is assigned for each area based on how aggressive the tumor appears. A tumor with cell that appear close to normal is assigned a low Gleason score (six or below). A tumor with cells that appear clearly different from those of a normal prostate is assigned a high Gleason score (seven or above). A system of grading prostate cancer tissue based on how it looks under a microscope. Gleason scores range from 2 to 10 and indicate how likely it is that a tumor will spread. A low Gleason score means the cancer tissue is similar to normal prostate tissue and the tumor is less likely to spread; a high Gleason score means the cancer tissue is very different from normal and the tumor is more likely to spread.
Time Frame: Baseline
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Treatment (Antihormone Therapy and Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 18
units on a scale | 8 [6 to 9]

3. Secondary Outcome: Levels of DHEA in Blood From Radical Prostatectomy Specimens
Time Frame: Up to 1 year
Measure: Median (95% Confidence Interval); unit: ng/dL
Arm/Group | Treatment (Antihormone Therapy and Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 18
ng/dL | 256 [81 to 461]

4. Secondary Outcome: Levels of DHEA-S in Blood From Radical Prostatectomy Specimens
Time Frame: Up to 1 year
Measure: Median (95% Confidence Interval); unit: mcg/dL
Arm/Group | Treatment (Antihormone Therapy and Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 18
mcg/dL | 90 [24.9 to 221]

5. Secondary Outcome: Levels of DHT in Blood From Radical Prostatectomy Specimens
Time Frame: Up to 1 year
Measure: Median (95% Confidence Interval); unit: ng/dL
Arm/Group | Treatment (Antihormone Therapy and Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 18
ng/dL | 24 [2 to 54]

6. Secondary Outcome: Levels of PSA in Blood From Radical Prostatectomy Specimens
Time Frame: Up to 1 year
Measure: Median (95% Confidence Interval); unit: ng/mL
Arm/Group | Treatment (Antihormone Therapy and Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 18
ng/mL | 9.44 [1.19 to 41.3]

7. Secondary Outcome: Levels of Testosterone in Blood From Radical Prostatectomy Specimens
Time Frame: Up to 1 year
Measure: Median (95% Confidence Interval); unit: ng/dL
Arm/Group | Treatment (Antihormone Therapy and Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 18
ng/dL | 319 [138 to 521]

8. Other Pre Specified Outcome: Protein Expression Analysis, Including AR Target Genes, PSA and TMPRSS2
Time Frame: Up to 1 year
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Safety and Tolerability of Androgen Depletion Therapy in Combination With Vorinostat as Assessed by Physical Examinations, Adverse Events, and Laboratory Assessments. Please See Adverse Events Section.
Description: Adverse events will be monitored at each scheduled visit and throughout the study. Toxicity will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Time Frame: Up to 1 year
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Gene Expression Analysis, Including AR Target Genes, PSA and TMPRSS2
Description: Estimates and 95% confidence intervals for the proportion of patients with nondetectable levels of PSA and TMPRSS2 will be computed.
Time Frame: at 12 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Gene Microarray Analysis
Time Frame: Up to 1 year
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Levels of Testosterone in Prostate Tissue
Time Frame: Up to 1 year
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Levels of DHT in Prostate Tissue
Time Frame: Up to 1 year
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Levels of Androstenediol in Prostate Tissue
Time Frame: Up to 1 year
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Levels of Androstenedione in Prostate Tissue
Time Frame: Up to 1 year
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Levels of DHEA in Prostate Tissue
Time Frame: Up to 1 year
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Levels of DHEA-S in Prostate Tissue
Time Frame: Up to 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 30 days after treatment
Arm/Group | Treatment (Antihormone Therapy and Enzyme Inhibitor Therapy)
Serious Adverse Events (participants affected / at risk) | 2/19
Other Adverse Events (participants affected / at risk) | 17/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Antihormone Therapy and Enzyme Inhibitor Therapy) (N=19)
Thrombosis (Cardiac disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Antihormone Therapy and Enzyme Inhibitor Therapy) (N=19)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 11 (24)
Blood bilirubin increased (Investigations) | 1 (1)
Cardiac disorders-Other, specify (Cardiac disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Creatinine increased (Investigations) | 2 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 11 (28)
Hypertension (Vascular disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 8 (20)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2)
INR increased (Investigations) | 2 (3)
Lymphocyte count decreased (Investigations) | 4 (6)
Neutrophil count decreased (Investigations) | 1 (1)
Pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less